CLINICAL TRIAL: NCT01090258
Title: Pilot Evaluation of Closed Loop Ventilation and Oxygen Controller
Acronym: CLOSER1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Professeur, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS-2009
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Cardiac Surgery; Mechanically Ventilated Patients
Keywords: cardiac surgery; mechanical ventilation; automation; weaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Automated settings (Experimental): Ventilator settings automatically adjusted by the evaluated system, concerning the FiO2, the respiratory rate, the inspiratory and expiratory pressures and related settings (triggers, pressurization ramp, inspiratory/expiratory time...)
  Interventions: Device: Hamilton ventilator (G5 modify to S1) Automated settings
- protocolized settings (Active Comparator): Ventilator settings performed by the local respiratory therapists according to the local protocols
  Interventions: Other: Hamilton ventilator (G5) protocolized settings

INTERVENTIONS:
Device: Hamilton ventilator (G5 modify to S1) Automated settings — Automated settings (respiratory rate [RR], FiO2, Insp and exp pressures) Ventilator settings automatically adjusted by the evaluated system, concerning the FiO2, the respiratory rate, the inspiratory and expiratory pressures and related settings (triggers, pressurization ramp, inspiratory/expiratory time...)
  Other Names: Intellivent
  Arms: Automated settings
Other: Hamilton ventilator (G5) protocolized settings — Mechanical ventilation settings performed by the respiratory therapists according to the local protocols
  Arms: protocolized settings

SUMMARY:
The study compares automated settings (Intellivent) with protocolized settings of the ventilator after cardiac surgery. The settings concern the respiratory rate, the inspiratory and expiratory pressure and FiO2. The aim of the study is to demonstrate that automated settings are feasible and safe.

The study design is a randomized controled study. 30 patients will be ventilated with automated mode and 30 patients with protocolized settings after cardiac surgery.

The hypothesis is that the automated mode allows a safer ventilation with better maintain of the patient in predefined optimal zone of ventilation.

DETAILED DESCRIPTION:
Aim: feasibility and safety study = evaluation of the possibility for a fully automated ventilator to safely manage the ventilation and oxygenation after cardiac surgery

Hypothesis:

Intellivent will maintain the patient with " optimal ventilation " better than during usual management with a minimal number of interventions

Monocentric: IUCPQ, Hôpital Laval, Québec Randomized controlled safety study, unblinded Patients after elective cardiac surgery Two arms Intellivent (fully automatic ventilation) Protocolized ventilation 4 hours study 60 patients planned to be included Primary outcome: number of episodes in the " not acceptable " zone of ventilation and duration

Secondary outcome:

Number of episodes in the " acceptable " zone of ventilation and duration Number of manual settings and duration of interventions Comparison of arterial blood gases Time to wean the FiO2 the PEEP Time to begin the assisted ventilation Duration of mechanical ventilation

ELIGIBILITY:
Criteria for consent (before surgical procedure):

* Elective cardiac surgery
* Age 18 to 90 years
* Absence of pregnancy
* Body Mass Index < 40 kg/m²
* Creatinine < 200micromol/L)
* Baseline PaCO2 > 50 mmHg)

Exclusion Criteria:

* Unexpected surgical procedure
* Major complication during surgery
* Early extubation expected (< 1 hour)
* Broncho-pleural fistula
* Study ventilator not available

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
" not acceptable " zone of ventilation | During the four hours of the study protocol
  Number of episodes, duration and percentage of time in the " not acceptable " zone of ventilation as pre-defined
" not acceptable " zone of ventilation | During the 4 hours of the protocol
  Number of episodes, duration and percentage of time in the " not acceptable " zone of ventilation as pre-defined

REFERENCES:
- [Derived] Lellouche F, Bouchard PA, Simard S, L'Her E, Wysocki M. Evaluation of fully automated ventilation: a randomized controlled study in post-cardiac surgery patients. Intensive Care Med. 2013 Mar;39(3):463-71. doi: 10.1007/s00134-012-2799-2. Epub 2013 Jan 22. PMID 23338569